CLINICAL TRIAL: NCT02405793
Title: A Phase 2b, Multicenter, Randomized, Single Blind, Fixed Dose, Parallel Group Study to Evaluate the Efficacy and Safety of Meloxicam SoluMatrix® [Test] Capsules and Meloxicam Tablets in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Brief Title: Meloxicam SoluMatrix® Capsules vs Meloxicam Tablets to Treat Osteoarthritis Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal business decision not to move forward with study
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEL2-14-05
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Meloxicam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meloxicam low dose test capsule (Experimental): Meloxicam SoluMatrix Capsules - low dose QD
  Interventions: Drug: Meloxicam Test Capsules
- Meloxicam high dose test capsule (Experimental): Meloxicam SoluMatrix Capsules - high dose QD
  Interventions: Drug: Meloxicam Test Capsules
- Meloxicam tablets (Active Comparator): Meloxicam Tablets QD
  Interventions: Drug: Meloxicam Tablets

INTERVENTIONS:
Drug: Meloxicam Test Capsules
  Arms: Meloxicam low dose test capsule
Drug: Meloxicam Test Capsules
  Arms: Meloxicam high dose test capsule
Drug: Meloxicam Tablets
  Arms: Meloxicam tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a low dose and a high dose of Meloxicam SoluMatrix® Capsules versus Meloxicam Tablets for the treatment of pain due to osteoarthritis of the knee or hip.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Functional Class I-III osteoarthritis (OA) of the hip or knee
* Chronic user of nonsteroidal anti-inflammatory drugs (NSAIDs) and/or acetaminophen for OA pain
* Discontinued all analgesic therapy at Screening
* For women of childbearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Ability to ambulate

Exclusion Criteria:

* History of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any NSAIDs, including meloxicam
* Requires regular (more than 2 doses per week) use of opioid or opioid combination products to control OA pain of the knee or hip
* Clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease
* Significant difficulties swallowing capsules/tablets or unable to tolerate oral medication
* Previous participation in another clinical study of Meloxicam Capsules or received any investigational drug or device or investigational therapy within 30 days before Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Pain Measured Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score. | Baseline to Week 6

SECONDARY OUTCOMES:
Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Function Measured Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score. | Baseline to Week 6
Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Stiffness Measured Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score. | Baseline to Week 6
Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Symptoms Measured Using the Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score. | Baseline to Week 6
Change From Pre-dose to 2 Hours Post-dose in Pain Intensity as Measured by the Numerical Pain Rating Scale on Day 3. | 2 hours after dosing on Day 3
Change From Pre-dose to 2 Hours Post-dose in Pain Intensity as Measured by the Numerical Pain Rating Scale on Day 14. | 2 hours after dosing on Day 14
Change From Pre-dose to 2 Hours Post-dose in Morning Stiffness Severity as Measured by the Numerical Rating Scale on Day 3. | 2 hours after dosing on Day 3
Change From Pre-dose to 2 Hours Post-dose in Morning Stiffness Severity as Measured by the Numerical Rating Scale on Day 14. | 2 hours after dosing on Day 14
Patient Global Impression of Change | Baseline to Week 6/Early Termination
Clinical Global Impression of Change | Baseline to Week 6/Early Termination
Amount of Rescue Medication Taken by Each Subject | Baseline to Week 6/Early Termination
Cumulative Discontinuations Due to Lack of Efficacy at Week 6 | Baseline to Week 6
Responders with at Least a 10-mm Improvement in Mean Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 6. | Baseline to Week 6
Safety of Meloxicam SoluMatrix Capsules low dose, Meloxicam SoluMatrix Capsules high dose, and Meloxicam Tablets as Assessed by the Incidence of Adverse Events From Baseline to Week 6 or Early Termination | Baseline to Week 6/Early Termination